CLINICAL TRIAL: NCT00885365
Title: A Multicentre, Multinational, Open-Label, Randomised, Parallel Group Clinical Trial of Tobrineb®/Actitob®/Bramitob® (Tobramycin Solution for Nebulisation, 300mg Twice Daily in 4mL Unit Dose Vials) Compared to TOBI® in the Treatment of Patients With Cystic Fibrosis and Chronic Infection With Pseudomonas Aeruginosa
Brief Title: A Study Comparing the Efficacy and Tolerability of Tobrineb®/Actitob®/Bramitob® Versus TOBI®
Acronym: CT03 Core
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMA-0631-PR-0010 Core
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-04

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; P. aeruginosa; tobramycin
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bramitob (Experimental): tobramycin / Bramitob administered 300mg twice a day for 4 weeks
  Interventions: Drug: tobramycin / Bramitob
- TOBI (Active Comparator): tobramycin / TOBI administered 300mg twice a day for 4 weeks
  Interventions: Drug: tobramycin / TOBI

INTERVENTIONS:
Drug: tobramycin / Bramitob — 300mg/4ml solution, via a nebuliser, over a 4-week treatment in a twice-daily regimen
  Other Names: Bramitob; Tobrineb; Actitob; Bethkis
  Arms: Bramitob
Drug: tobramycin / TOBI — 300mg/5ml solution administered via nebuliser, over a 4-week treatment in a twice-daily regimen
  Other Names: TOBI
  Arms: TOBI

SUMMARY:
The objectives of the study are to demonstrate that Tobrineb®/Actitob®/Bramitob® is non-inferior to TOBI® in the primary efficacy variable, forced expiratory volume in one second (FEV1) percent of predicted normal, and to compare the safety in participants with cystic fibrosis and chronic infection of the lungs with Pseudomonas aeruginosa.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged ≥ 6;
* Clinical diagnosis of cystic fibrosis defined as: (1)Patients preferably registered in the National Registry of CF (or other documents depending on country legislation); (2) Evidence of two or more typical pulmonary clinical features observed in CF, e.g., persistent colonization/infection with typical CF pathogens, chronic cough and sputum production, persistent chest radiography abnormalities, airway obstruction, nasal polyps and/or digital clubbing;
* Positive response in the standard sweat test (sweat chloride concentration ≥ 60 mmol/l for the standard method or ≥ 80 mmol/L for a microduct technique) documented in the clinical records and/or gene mutation documented in the clinical records;
* Chronic colonization of P. aeruginosa: presence in a sputum or throat culture of a minimum of 2 positive samples for P. aeruginosa over the previous 12 months and/or presence of more than two precipitating antibodies against P. aeruginosa;
* Sputum containing P. aeruginosa susceptible to tobramycin (defined as a zone diameter ≥ 16 mm after testing with 10 µg tobramycin disk or as a minimal inhibition concentration based on microdilution testing system) as identified by local laboratory at screening visit;
* Forced expiratory volume in 1 sec (FEV₁) ≥ 40% and ≤ 80% of the predicted normal value;
* Written informed consent obtained by parents/legal representative according to local regulations) and by the patient (when appropriate).

Exclusion Criteria:

* Administration of antipseudomonal antibiotic therapy by any route in the previous 4 weeks;
* Evidence of impaired renal function (serum creatinine level ≥ 1.5 mg/dl);
* Evidence of impaired auditory function (auditory threshold in either ear above 20 dB at frequencies between 250 and 8000Hz);
* Sputum culture containing Burkholderia cepacia;
* Patients with end-stage lung disease, candidates for heart-lung transplantation;
* History of other clinically significant cardiac, renal, neurological, gastrointestinal, hepatic or endocrine disease related to cystic fibrosis, whose sequelae and/or treatment can interfere with the results of the present study;
* Female subjects: pregnant or with active desire to be pregnant, lactating mother or lack of efficient contraception in a subject with child-bearing potential (i.e., contraceptive methods other than rod containing a hormone that prevents user from getting pregnant and that will be placed under the skin, syringes that contain a contraceptive hormone, combined birth control pill, i.e., such that contains two hormones, some intrauterine devices (IUDs) and sexual abstinence). A pregnancy test in urine is to be carried out in women of a fertile age at screening and at the last clinic visit;
* Known hypersensitivity to aminoglycosides;
* Patients with evidence of alcohol or drug abuse, likely to be not compliant with the study protocol or likely to be not compliant with the study treatments;
* Participation in another clinical trial with an investigational drug in the four weeks preceding the screening visit.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henryk Mazurek, Doctor, Principal Investigator — Klinika Pneumonologii i Mukowiscydozy, Instytut Gruzlicy i Chorob Pluc w Rabce Zdroj
Locations (44):
- Centrum pro cystickou fibrosu, Pediatricka klinika UK 2.LF, Fakultní nemocnice v Motole, Prague, Czechia
- France (3):
  - CHR Clemenceau, Caen
  - Hopital Arnaud de Villeneuve, Clinique des maladies respiratoires, Montpellier
  - Hopital Necker, Paris
- Germany (2):
  - Pädiatrische Pneumologie und Allergologie, Mukovizidose-Zentrum, Zentrum für Kinderheilkunde und Jugendmedizin, GieBen
  - HELIOS Klinikum Krefeld, Zentrum für Kinder- und Jugendmedizin, Krefeld
- Hungary (3):
  - Fővárosi Önkormányzat Heim Pál, Budapest
  - Kaposi Mór Oktatókórház, Mosdós
  - Szegedi Tudományegyetem Szent-Györgyi Albert Orvos- és Gyógyszerésztudományi Centrum, Szeged
- Poland (9):
  - Specjalistyczny ZOZ nad Matka i Dzieckiem, Poradnia Leczenia Mukowiscydozy, Gdansk
  - I Oddzial Chorob Dzieciecych, Wojewodzki Specjalistyczny Szpital Dzieciecy, Kielce
  - Oddzial Kliniczny Interny Dzieciecej i Alergologii, Wojewodzki Szpital Specjalistyczny, Lodz
  - Dzieciecy Szpital Kliniczny Akademii Medycznej, Klinika Chorob Pluc I Reumatologii, Lublin
  - Multiple Locations
  - Klinika Pneumonologii, Alergologii Dzieciecej i Immunologii Klinicznej Szpital Kliniczny Uniwersytetu Medycznego w Poznaniu, Poznan
  - Klinika Pneumonologii i Mukowiscydozy, Instytut Gruzlicy i Chorob Pluc w Rabce Zdroj, Rabka-Zdrój
  - Poradnia Mukowiscydozy Wojewodzkiej, Przychodni Specjalistycznej dla Dzieci, Szpitala Wojewodzkiego Nr 2, Rzeszów
  - Klinika Pediatrii Instytut Matki I Dziecka, Warsaw
- Russia (10):
  - State Medical Institution: Republican Childrens Clinical Hospital under the Ministry of Health of the Republic of Tatarstan, Kazan'
  - Federal State Institution: Scientific Research Pulmonology Institute under the Roszdrav, Moscow
  - State Medical Institution: Filatov Chidren's City Clinical Hospital #13, Moscow
  - Federal State Institution "Nizhegorodskiy Research Institute of Children's Gastroenterology of Russian Medical Technologies", Nizhny Novgorod
  - State Medical Institution: Regional Children's Hospital Pulmonology Department, Rostov-on-Don
  - Saint-Petersburg State Medical Institution: City Children's Hospital of Saint Olga, Saint Petersburg
  - Regional State Medical Institution: Smolensk Regional Children's Clinical Hospital, Smolensk
  - State Higher Educational Institution: Bashkir State Medical University under the Roszdrav, Ufa
  - State Higher Educational Institution: Burdenko Voronezh State Medical Academy under the Roszdrav, Voronezh
  - Minicipal Medical Institution: Children's Clinical Hospital #1, Yaroslavl
- Spain (7):
  - Complejo Hospitalario Universitario A Coruña (Hospital Materno-Infantil Teresa Herrera), A Coruña
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario La Paz, Madrid
  - Corporació Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Ntra Sra. De la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario La Fe, Valencia
  - Hospital Universitario Miguel Servet (Children), Zaragoza
- Ukraine (9):
  - Dnipropetrovsk City Children Clinical Hospital # 2, Dnipropetrovsk
  - Donetsk Regional Children Clinical Hospital, Donetsk
  - Kriviy Rig City Clinical Hospital # 8, Kryvyi Rih
  - Institute of Phthysiology and Pulmonology n.a., F.G.Yanovskiy of the Academy of Medical Science of Ukraine, Kyiv
  - Institute of Pediatrics, Obstetrics and Gynecology of the Academy of Medical Science of Ukraine, Kyiv
  - Lviv Regional Children Specialized Clinical Hospital, Lviv
  - Odesa Regional Children Clinical Hospital, Odesa
  - Simferopol Central District Clinical Hospital, Simferopol
  - Zaporizhya Regional Clinical Children Hospital, Zaporizhya

REFERENCES:
- [Result] Mazurek H, Chiron R, Kucerova T, Geidel C, Bolbas K, Chuchalin A, Blanco-Aparicio M, Santoro D, Varoli G, Zibellini M, Cicirello HG, Antipkin YG. Long-term efficacy and safety of aerosolized tobramycin 300 mg/4 ml in cystic fibrosis. Pediatr Pulmonol. 2014 Nov;49(11):1076-89. doi: 10.1002/ppul.22989. Epub 2014 Jan 24. PMID 24464974
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=CMA-0631-PR-0010

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 406 participants screened, 324 participants randomized
Period: 4 Weeks ON Treatment
Arm/Group | Bramitob | TOBI
Started | 159 | 165
Intent-to-Treat Population | 158 (Participants who took 1 dose of study medication and had baseline and at least 1 post-treatment FEV1) | 163
Safety Population | 156 (Nine participants randomized to Bramitob were administered TOBI.) | 168 (Six participants randomized to TOBI were administered Bramitob)
Completed | 155 | 159
Not Completed | 4 | 6
Not completed — Adverse Event | 2 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Period: 4 Weeks OFF Treatment
Arm/Group | Bramitob | TOBI
Started | 155 | 159
Completed | 155 | 159
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Bramitob | TOBI | Total
Number analyzed (Participants) | 156 | 168 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.95 (6.74) | 15.74 (7.24) | 15.84 (6.99)
Age, Customized [Number; unit: participants]
  6-12 years | 49 | 54 | 103
  13-17 years | 50 | 62 | 112
  > 17 years | 57 | 52 | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 83 | 167
  Male | 72 | 85 | 157
Race/Ethnicity, Customized [Number; unit: participants]
  White | 156 | 168 | 324
Height [Mean (Standard Deviation); unit: centimeters] | 153.05 (17.31) | 153.41 (19.88) | 153.24 (18.66)
Weight [Mean (Standard Deviation); unit: kilograms] | 42.64 (14.92) | 43.81 (16.39) | 43.25 (15.69)
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meters^2] | 17.55 (3.12) | 17.79 (3.32) | 17.68 (3.22)
Time from diagnosis of chronic colonization of P. aeruginosa [Mean (Standard Deviation); unit: years] | 2.27 (4.22) | 2.36 (4.23) | 2.31 (4.22)
Time from first Cystic Fibrosis diagnosis [Mean (Standard Deviation); unit: years] | 12.16 (6.13) | 11.74 (6.55) | 11.94 (6.34)
Tobramycin Minimal Inhibitory Concentration (MIC) value [Number; unit: participants] — MIC is the lowest concentration of tobramycin that completely inhibits visible growth of a micro-organism.
  participants
    <16 mcg/mL | 143 | 159 | 302
    >=16 mcg/mL | 13 | 8 | 21
    Missing | 0 | 1 | 1
Forced Expiratory Volume in 1 second (FEV1) [Number; unit: participants]
  <50 % predicted | 37 | 38 | 75
  >=50 % predicted | 119 | 130 | 249
Use of rhDNase [Number; unit: participants] — Baseline use of rhDNase is set to 'Yes' if a patient has used rhDNase on the same date or within the 10 days prior to start of study drug administration. If the timing of rhDNase use cannot be identified because of missing date, then the use of rhDNase at baseline is considered as 'Yes'.
  participants
    Yes | 110 | 119 | 229
    No | 46 | 49 | 95

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of the Treatment Period of Forced Expiratory Volume in 1 Second (FEV1), Expressed as Percentage of Predicted Normal
Description: Pulmonary function measurements were performed by using a self-calibrated computer-operated pneumotochographic spirometer at all clinic visits. Because this study included both adults and children and lung volume is an age-dependent variable, reference normal FEV1 values for children were different than the reference normal values used with adult participants. Three measurements were collected and the greatest FEV1 value was recorded.
Time Frame: Day 0 (baseline), Week 4
Population: Intent-to-Treat (ITT) Population, Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: percentage predicted FEV1
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 158 | 163
percentage predicted FEV1 | 6.99 (9.52) | 7.51 (9.63)
Statistical Analysis 1: Comparison: Bramitob vs TOBI; Based on previous studies, the difference between reference and placebo after 4-week treatment is assumed to be about 12% and the non-inferiority margin safely placed at 4.5%. With a between-patient SD of 13.5% and estimated difference between treatments of zero, sample size of 143 per group allows a 80% power to show the non-inferiority of Bramitob® versus TOBI®. Accounting for an expected dropout rate of 11%, a minimum of 160 participants per group is required; Test type: Non-Inferiority or Equivalence — The non-inferiority is shown if the lower limit of the two-sided 95% confidence interval is above the non-inferiority margin set at -4.5%; p = 0.640, ANCOVA; difference of least square means = -0.50, 95% CI 2-sided [-2.58 to 1.59]

2. Secondary Outcome: Change From Baseline to End of Weeks 2, 4, and 8 of Forced Expiratory Volume in 1 Second (FEV1), Expressed as Percentage of Predicted Normal
Description: Pulmonary function measurements were performed by using a self-calibrated computer-operated pneumotochographic spirometer at all clinic visits. Because this study included both adults and children and lung volume is an age-dependent variable, reference normal FEV1 values for children were different than the reference normal values used with adult participants. Three measurements were collected and the greatest FEV1 value was recorded. Observed values are summarized (without last observation carry forward).
Time Frame: Day 0 (baseline), Week 2, Week 4, Week 8
Population: Intent-to-Treat (ITT) Population, observed values. Differences in number of participants analyzed to the ITT population represent participants who missed visits, or failed to take the FEV1 test.
Measure: Mean (Standard Deviation); unit: percentage predicted FEV1
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 158 | 163
percentage predicted FEV1
  Week 2 [n=158, 163] | 6.70 (9.99) | 6.93 (9.40)
  Week 4 [N=155, 161] | 7.10 (9.57) | 7.63 (9.61)
  Week 8 [n=155, 159] | 5.47 (11.88) | 5.37 (11.11)

3. Secondary Outcome: Change From Baseline to End of Weeks 2, 4, and 8 of Absolute Forced Expiratory Volume in 1 Second (FEV1)
Description: Pulmonary function measurements were performed by using a self-calibrated computer-operated pneumotochographic spirometer at all clinic visits. Three measurements were collected and the greatest FEV1 value was recorded. Observed values are summarized (without last observation carry forward).
Time Frame: Day 0 (baseline), Week 2, Week 4, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 158 | 163
liters
  Week 2 [n=158, 163] | 0.18 (0.27) | 0.19 (0.27)
  Week 4 [n=155, 161] | 0.20 (0.29) | 0.22 (0.28)
  Week 8 [n=155,159] | 0.16 (0.33) | 0.16 (0.32)
Statistical Analysis 1: Comparison: Bramitob vs TOBI; Analysis for Week 4; Test type: Superiority or Other; p = 0.634, ANCOVA; difference of least square means = -0.01, 95% CI 2-sided [-0.08 to 0.05]

4. Secondary Outcome: Change From Baseline at End of Weeks 2, 4, and 8 of Forced Vital Capacity (FVC) Expressed as Percentage of Predicted Normal
Description: FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. It is measured via spirometry. Because this study included both adults and children and lung volume is an age-dependent variable, reference normal FVC values for children were different than the reference normal values used with adult participants.
Time Frame: Day 0 (baseline), Week 2, Week 4, Week 8
Population: Intent-to-Treat (ITT) Population, observed values. Differences in number of participants analyzed to the ITT population represent participants who missed visits, or failed to take the FVC test.
Measure: Mean (Standard Deviation); unit: percentage predicted FVC
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 156 | 163
percentage predicted FVC
  Week 2 [n=156, 163] | 4.36 (10.81) | 5.36 (10.03)
  Week 4 [n=153, 161] | 4.83 (10.05) | 5.58 (10.86)
  Week 8 [n=153,159] | 2.70 (12.30) | 5.04 (12.21)
Statistical Analysis 1: Comparison: Bramitob vs TOBI; Analysis for Week 4; Test type: Superiority or Other; p = 0.630, ANCOVA; difference of least square means = -0.55, 95% CI 2-sided [-2.78 to 1.69]

5. Secondary Outcome: Change From Baseline to End of Weeks 2, 4, and 8 of Absolute Forced Vital Capacity (FVC)
Description: FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. It is measured via spirometry.
Time Frame: Day 0 (baseline), Week 2, Week 4, Week 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 156 | 163
liters
  Week 2 [n=156, 163] | 0.14 (0.34) | 0.16 (0.32)
  Week 4 [n=153, 161] | 0.16 (0.34) | 0.18 (0.36)
  Week 8 [n=153,159] | 0.10 (0.38) | 0.16 (0.39)
Statistical Analysis 1: Comparison: Bramitob vs TOBI; Analysis for Week 4; Test type: Superiority or Other; p = 0.693, ANCOVA; difference of least square means = -0.02, 95% CI 2-sided [-0.09 to 0.06]

6. Secondary Outcome: Change From Baseline to End of Weeks 2, 4, and 8 of Forced Expiratory Flow at 25-75% of Vital Capacity (FEF 25-75%), Expressed as Percentage of Predicted Normal
Description: Difference in the forced expiratory flow rate in mid-exhalation as a percent of predicted to standard values measured from baseline to weeks 2 (treated), 4 (treated), and 8 (untreated). Because this study included both adults and children and lung volume is an age-dependent variable, reference normal FEF 25-75% values for children were different than the reference normal values used with adult participants.
Time Frame: Day 0 (baseline), Week 2, Week 4, Week 8
Population: Intent-to-Treat (ITT) Population, observed values. Differences in number of participants analyzed to the ITT population represent participants who missed visits, or failed to take the FEF 25-75% test.
Measure: Mean (Standard Deviation); unit: percentage predicted FEF 25-75%
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 156 | 162
percentage predicted FEF 25-75%
  Week 2 [n=156, 162] | 10.30 (17.07) | 8.57 (19.00)
  Week 4 [n=154, 159] | 10.44 (15.17) | 9.32 (17.99)
  Week 8 [n=154,158] | 9.05 (19.59) | 6.41 (20.46)
Statistical Analysis 1: Comparison: Bramitob vs TOBI; Analysis for Week 4; Test type: Superiority or Other; p = 0.777, ANCOVA; difference of least square means = 0.51, 95% CI 2-sided [-3.06 to 4.09]

7. Secondary Outcome: Change From Baseline to End of Weeks 2, 4, and 8 of Forced Expiratory Flow at 25-75% of Vital Capacity (FEF 25-75%)
Description: Difference in the forced expiratory flow rate in mid-exhalation measured from baseline to weeks 2 (treated), 4 (treated), and 8 (untreated).
Time Frame: Day 0 (baseline), Week 2, Week 4, Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liters/second
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 156 | 162
liters/second
  Week 2 [n=156, 162] | 0.32 (0.50) | 0.28 (0.56)
  Week 4 [n=154, 159] | 0.34 (0.48) | 0.29 (0.57)
  Week 8 [n=154,158] | 0.28 (0.57) | 0.21 (0.67)
Statistical Analysis 1: Comparison: Bramitob vs TOBI; Analysis for Week 4; Test type: Superiority or Other; p = 0.505, ANCOVA; difference of least square means = 0.04, 95% CI 2-sided [-0.08 to 0.15]

8. Secondary Outcome: Change From Baseline to End of Weeks 4 and 8 in Pseudomonas Aeruginosa Log10 Bacterial Load in Sputum
Description: If a participant had more than one Pseudomonas aeruginosa (PA) morphotype at a given visit, and therefore more than one bacterial load value, then the bacterial load value corresponding to the highest tobramycin minimal inhibitory concentration (MIC) value regardless of the PA morphotype was used. If the tobramycin MIC value was the same for different PA morphotypes, then the bacterial load value corresponding to morphotype 1 (mucoid colony) was used. If morphotype 1 was not available, bacterial load value corresponding to morphotype 2 (dry colony) was used.
Time Frame: Day -10 to -1 (baseline), Week 4, Week 8
Population: Intent-to-Treat (ITT) Population; At Week 4, six Bramitob patients and seven TOBI patients were missing sputum samples. At Week 8, 11 Bramitob patients and 16 TOBI patients were missing sputum samples.
Measure: Mean (Standard Deviation); unit: colony forming units/gram
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 158 | 163
colony forming units/gram
  Week 4 [n=152, 156] | -2.14 (2.41) | -2.07 (2.20)
  Week 8 [n=147, 147] | -0.72 (2.17) | -0.87 (2.23)
Statistical Analysis 1: Comparison: Bramitob vs TOBI; Analysis of Week 4 data; Test type: Superiority or Other; p = 0.820, ANCOVA — A priori threshold for statistical significance is <= 0.050; treatment and country are fixed effects and baseline log10 bacterial load (CFU/g) value is a covariate; difference of least square means = 0.04, 95% CI 2-sided [-0.31 to 0.39], Standard Error of Mean 0.18

9. Secondary Outcome: Minimal Inhibitory Concentration Inhibiting Growth of 50% (MIC50) of Pseudomonas Aeruginosa
Description: MIC50 is the concentration of tobramycin required to inhibit 50% of Pseudomonas aeruginosa. MIC values were calculated for three different Pseudomonas aeruginosa (PA) strains:
  * Morphotype 1: mucoid
  * Morphotype 2: dry
  * Morphotype 3: variant
  Overall MIC50 values are reported. If a participant has more than one PA morphotype at a given visit, then the highest tobramycin MIC value was used, regardless of PA morphotype. If a participant has more than one available result for each morphotype then the highest tobramycin MIC value was used. If the tobramycin MIC values are equal then the MIC value for the isolate with the highest bacterial load value was used.
Time Frame: Week 4, Week 8
Population: Intent-to-Treat (ITT) Population
Measure: Number; unit: micrograms/milliliters
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 158 | 163
micrograms/milliliters
  Week 4 [n=126, 134] | 1 | 0.5
  Week 8 [n=129, 128] | 1 | 1

10. Secondary Outcome: Minimal Inhibitory Concentration Inhibiting Growth of 90% (MIC90) of Pseudomonas Aeruginosa
Description: MIC90 is the concentration of tobramycin required to inhibit 90% of Pseudomonas aeruginosa. MIC values were calculated for three different Pseudomonas aeruginosa (PA) strains:
  * Morphotype 1: mucoid
  * Morphotype 2: dry
  * Morphotype 3: variant
  Overall MIC90 values are reported. If a participant has more than one PA morphotype at a given visit, then the highest tobramycin MIC value was used, regardless of PA morphotype. If a participant has more than one available result for each morphotype then the highest tobramycin MIC value was used. If the tobramycin MIC values are equal then the MIC value for the isolate with the highest bacterial load value was used.
Time Frame: Week 4, Week 8
Population: Intent-to-Treat (ITT) Population
Measure: Number; unit: micrograms/milliliters
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 158 | 163
micrograms/milliliters
  Week 4 [n=126, 134] | 32 | 32
  Week 8 [n=129, 128] | 32 | 32

11. Secondary Outcome: Microbiological Outcome Summary by Visit
Description: Microbiological outcomes are derived considering all P. aeruginosa (PA) morphotypes together.
  Week 4 and Week 8 microbiological outcomes:
  * Eradication = elimination of PA
  * Persistence = persistence of PA detected at previous visit
  * Superinfection = appearance of a pathogen (other than PA) not detected at previous visit
  * Re-infection (week 8 only) = re-appearance of PA detected at Screening and eradicated at Week 4
  Superinfection supersedes eradication. Persistence for P. aeruginosa supersedes superinfection.
  Re-infection for P. aeruginosa supersedes superinfection.
Time Frame: Day -10 to -1 (screening), Weeks 4 and 8
Population: Intent-to-Treat Population.
Measure: Number; unit: percentage of participants
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 158 | 163
percentage of participants
  Screening: Presence of P aeruginosa | 100 | 100
  Week 4: Eradication | 9.2 | 7.1
  Week 4: Persistence | 82.9 | 85.3
  Week 4: Superinfection | 7.9 | 7.7
  Week 8: Eradication | 2.7 | 3.4
  Week 8: Persistence | 78.9 | 83.0
  Week 8: Superinfection | 9.5 | 9.5
  Week 8: Re-infection | 8.8 | 4.1
Statistical Analysis 1: Comparison: Bramitob vs TOBI; Week 4; Test type: Superiority or Other; p = 0.692, Cochran-Mantel-Haenszel — A priori threshold for statistical significance is <= 0.050; Test controlling for country
Statistical Analysis 2: Comparison: Bramitob vs TOBI; Week 8; Test type: Superiority or Other; p = 0.128, Cochran-Mantel-Haenszel — A priori threshold for statistical significance is <= 0.050; Test controlling for country

12. Secondary Outcome: Change From Baseline to End of Weeks 2, 4 and 8 in Body Weight
Description: Body weight was measured at all study visits as part of the physical examination.
Time Frame: Day 0 (baseline), Weeks 2, 4 and 8
Population: Intent-to-Treat (ITT) Population, observed values. Two participants from both treatment arms were missing data at Week 4. Three participants from Bramitob and 4 participants from TOBI were missing data at Week 8.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 158 | 163
kilograms
  Week 2 [n=158, 163] | 0.24 (0.68) | 0.22 (0.72)
  Week 4 [n=156, 161] | 0.39 (0.90) | 0.42 (0.97)
  Week 8 [n=155,159] | 0.60 (1.14) | 0.53 (1.27)

13. Secondary Outcome: Change From Baseline to End of Weeks 2, 4 and 8 in Body Mass Index (BMI)
Time Frame: Day 0 (baseline), Weeks 2, 4 and 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kilograms/meters^2
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 158 | 163
kilograms/meters^2
  Week 2 [n=158, 163] | 0.10 (0.28) | 0.10 (0.29)
  Week 4 [n=156, 161] | 0.12 (0.37) | 0.13 (0.38)
  Week 8 [n=155,159] | 0.16 (0.48) | 0.14 (0.49)

14. Secondary Outcome: Count of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-Emergent Adverse Events defined as adverse events occurring after the first intake of study treatment (or the same day).
  The investigator assessed relation to study treatment as a binary question: Reasonable possibility of relatedness or no reasonable possibility of relatedness. The expression "reasonable possibility of relatedness" is meant to convey in general that there are facts (evidence) or arguments meant to suggest a causal relationship.
  A serious AE results in death, is life-threatening, requires hospitalization or prolongation of existing inpatient hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or an important medical event.
  The investigator rates the severity of the AE based on a three point scale: mild, moderate or severe. A severe event prevents any usual routine activity of the participant and causes severe discomfort.
Time Frame: Day 0 to Week 8
Population: Safety population: all randomised patients who took at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 156 | 168
percentage of participants
  TEAE | 31.4 | 28.0
  Related TEAE | 6.4 | 6.0
  Serious TEAE | 3.8 | 1.2
  Severe TEAE | 1.9 | 1.2
  TEAE leading to withdrawal | 0.6 | 3.0

15. Secondary Outcome: Participants With a Hearing Threshold >20 Decibel in at Least One Ear
Description: The potential ototoxic effects (hearing loss) of tobramycin were investigated by performing audiometric tests. Participants with a loss of auditory acuity greater than the 20 decibels auditory threshold are reported.
Time Frame: Day -10 to -1 (screening), Weeks 4 and 8
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Bramitob | TOBI
Number analyzed (Participants) | 156 | 168
percentage of participants
  Screening | 0 | 0
  Week 4 | 1.9 | 1.2
  Week 8 | 1.3 | 1.2

ADVERSE EVENTS:
Time Frame: Day 0 to Week 8
Arm/Group | Bramitob | TOBI
Serious Adverse Events (participants affected / at risk) | 6/156 | 2/168
Other Adverse Events (participants affected / at risk) | 10/156 | 10/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bramitob (N=156) | TOBI (N=168)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bramitob (N=156) | TOBI (N=168)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon PI submission of publication to Sponsor, Sponsor will complete its review within 90 days after receipt. At Sponsor's request, publication may be delayed up to 120 additional days for Sponsor to file necessary patent applications. In multicenter trials, PIs will postpone single center publications until after multicenter data publication. If no multicenter publication occurs within 12 months of trial completion, PI may publish single center results, subject to review timelines listed above.